CLINICAL TRIAL: NCT02704247
Title: Evaluation of CARDIOSPACE System in Healthy Volunteers for Physiological Research in Space Environment
Brief Title: CARDIOSPACE Evaluation in Healthy Volunteers
Acronym: CARDIOSPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: National Center for Spatial Study, Toulouse (Unknown); Astronaut Center of China (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHU-P 2014-01
Record Dates: First submitted 2014-06-04; First posted 2016-03-09 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Testing CARDIOSPACE System (Experimental): Healthy volunteers have to test CARDIOSPACE System
  Interventions: Device: CARDIOSPACE System

INTERVENTIONS:
Device: CARDIOSPACE System — * autonomic nervous system test
  * tilt test
  * ultrasound exploration at rest (heart / vessels)
  * laser doppler + iontophoresis test
  * sub-maximal exercise test
  Other Names: Physiological tests

SUMMARY:
The aim of this porject is to test the Cardiospace system that integrates several medical devices to monitor the cardiovascular system:

* ECG
* Brachial blood pressure
* Continuous finger blood pressure
* Ultrasound
* Laser doppler + iontophoresis Cardiospace will be used in space station to monitor the cardiovascular system of astronauts for research purpuse.

ELIGIBILITY:
Inclusion Criteria:

* Age : 18 to 40 years
* Size : 160 à 180
* Weight : BMI between 18 and 24
* Medical history :

  * No history of cardiovascular disease
  * No chronic treatment
  * No syncopal events (>2 by year)
* Physical examination

  * Normal cardio-pulmonary ausculation
  * Normal (DBP [60 - 90] SBP [100 - 140]
  * Normal heart rate (between 50 and 80 at rest)
* Complementary examination

  * Normal Electrocardiogram
  * Presence of temporal acoustic window
* Capable to understand the objectives and constraints of this study
* Covered by health social insurance
* Have signed the informed consent

Exclusion Criteria:

* Pregnant woman (beta HCG by urinary test) or breastfeeding

  * Refusing to sign the informed consent
  * Don't understand the objectives of this study
  * Minors or majors protect by the law
  * Don't Benefit of social insurance
  * Participation at the time of study enrolment during the present trial period in another clinical trial investigating.
  * Having reached or surpassed the annual amount of compensation allowed by clinical trials
  * Receipt of any chronic and regular treatment
  * Presence of sign cardiovascular diseases during the questioning
  * Presence of sign cardiovascular diseases during the examination
  * Presence of sign syncopals events ATCD diseases during the questioning (>2 by year)
  * Absence of temporal acoustic window with the Transcranial Doppler
  * Respiratory disorder, asthma
  * Any troubles preventing the realization of physical activity

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Heart rate measure on ECG | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine CUSTAUD, MD, PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Centre de Recherche Clinique, CHU d'Angers, Angers, France

IPD SHARING:
Plan to Share IPD: No